CLINICAL TRIAL: NCT03466541
Title: Workplace Interventions Preventing Risky Use of Alcohol and Sick Leave
Acronym: WIRUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Stavanger (Other)
Collaborators: Kompetansesenter rus - region vest Stavanger (KoRus) (Unknown); Stamina Helse (Unknown); Presenter (Unknown); University of Oslo (Other); Oslo Metropolitan University (Other); Alcohol and Drug Research Western Norway (KoRFor) (Unknown); Norwegian Institute of Public Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AA0000
Record Dates: First submitted 2018-03-08; First posted 2018-03-15 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Alcohol Consumption; Sick Leave; Workplace Interventions; Presenteeism
Keywords: Alcohol consumption; Sick leave; Workplace interventions; Presenteeism
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Riskbruk (Experimental): The employees randomised to the Riskbruk group will be offered two consultations a ∼15 min with the OHS. The subjects will receive individual feedback on the screening results. During these sessions, Motivational Interviewing will be used.
  Interventions: Behavioral: Riskbruk
- Balance (Experimental): The group allocated to the Balance intervention will follow a comprehensive multi-session eHealth intervention with personalised feedback on the screening results.
  Interventions: Behavioral: Balance
- Control group/usual care (No Intervention): The control group will receive the usual follow-up provided by the OHS for persons with risky alcohol behaviour. In order to provide something that appears as a plausible follow-up to the control participants, they will be given a booklet that covers general information about alcohol and potential risks and harms of drinking. The booklet contains no advise on how to achieve a change in drinking behaviour.

INTERVENTIONS:
Behavioral: Riskbruk — The Riskbruk model incorporates alcohol screening through a widely employed alcohol screening questionnaire, the Alcohol Use Disorders Identification Test (AUDIT) and a standard alcohol biomarker, carbohydrate-deficient transferring in serum (CDT), with brief consultations using the motivational interviewing (MI) technique. MI is a collaborative conversation style used to increase awareness and reflection around one's own drinking habits, as well as strengthening the person's motivation for a lifestyle change. The conversation style includes expressing empathy through reflective listening, communicating respect and acceptance of the participants and their feelings, and open up for self-reflection and exploration around the drinking behaviour.
  Arms: Riskbruk
Behavioral: Balance — Balance is a new Norwegian eHealth programme, and incorporates two approaches to behaviour modification interventions: a brief interventions and an intensive self-help programme. The intervention is based on cognitive-behavioural and self-help principles, and is given to the participants through multiple interactive sessions.
  Arms: Balance

SUMMARY:
The aim of this study is to investigate the effectiveness of two workplace interventions (the Riskbruk model and Balance) in reducing risky alcohol consumption, sickness absence and presenteeism. The purpose is to assess whether the Riskbruk model should be implemented in the Norwegian workforce in its entirety, whether the less extensive and costly alternative Balance is sufficient, or if neither one of them show effectiveness compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Employees screening positive for at-risk drinking (8+ on the AUDIT)

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2013-08; Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in alcohol consumption | Baseline and 6 months
Change in sickness absence | Baseline and 6 months

SECONDARY OUTCOMES:
Change in presenteeism | Baseline and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Stavanger, Stavanger, Rogaland, Norway